CLINICAL TRIAL: NCT05812768
Title: Suture-Tight™ First-in-Human Safety and Performance Study (CLP-05)
Brief Title: Suture-Tight™ First-in-Human Safety and Performance Study
Acronym: Suture-Tight™
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Vesteck, Inc. (Industry)
Collaborators: Prince of Wales Hospital, Sydney (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CLP-05
Record Dates: First submitted 2023-03-27; First posted 2023-04-14 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2023-03

CONDITIONS: Aortic Aneurysm, Abdominal
Keywords: EVAR; AAA; Anchor
MeSH Terms: conditions — Aortic Aneurysm, Abdominal

STUDY DESIGN:
Intervention Model Description: Subjects meeting all inclusion/exclusion criteria and scheduled for an EVAR procedure.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Suture-Tight (Experimental): Subjects meeting all inclusion and exclusion criteria will receive graft anchoring utilizing the Suture-Tight Suture Delivery System.
  Interventions: Device: Suture-Tight Suture Delivery System

INTERVENTIONS:
Device: Suture-Tight Suture Delivery System — Implantation of the Suture-Tight Suture in the deployment of multiple nitinol sutures to provide augmented fixation and sealing between endovascular aortic graft and the native artery.

SUMMARY:
Single center, open label, prospective, single-arm, first-in-human (FIH), pre-market clinical study with the objective of validating the safety and performance of the Suture-Tight™ Suture Delivery System in an EVAR procedure.

DETAILED DESCRIPTION:
Single center, study conducted at the Prince of Wales Private Hospital in Randwick, Australia. Up to 6 subjects may be enrolled. 1 to 3 subjects will complete initial enrollment and be followed for 30-days evaluating procedure and device safety. Additional subjects may be enrolled following the safety review to complete the 6-subject study. All subjects will be followed for six (6) months.

Subjects meeting all inclusion and exclusion criteria will be consented to receive an elective endovascular aortic aneurysm repair (EVAR) with graft anchoring utilizing the Suture-Tight device. Procedure and device safety and performance will be evaluated at 1- and 6-months by completing CT scans and KUB x-rays.

Data may be used to support a pivotal study of the investigational device and future global regulatory submissions.

ELIGIBILITY:
Inclusion Criteria:

* Currently scheduled for an elective endovascular repair of an abdominal aortic aneurysm (AAA) by EVAR with CT scan from within last 4 months. Acceptable AAA parameters include: AAA ≥ 5.0 cm in diameter OR AAA ≥ 4.5 cm in diameter with an increase of ≥ 0.5 cm within the past 6-months or ≥ 1.0 cm over the past 12-months
* Neck diameter, length and angulation that meets labeling requirements for the endograft used
* Successful EVAR graft placement with no evidence of EVAR-associated serious adverse event.

Exclusion Criteria:

* Mycotic or inflammatory AAA
* Prior surgical repair of an AAA
* Renal dialysis or significant chronic renal failure
* Evidence of recent acute coronary disease, thrombotic disease, or cerebral infarct
* Pregnancy

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2023-12-12 (Actual); Primary Completion 2024-07-19 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Serious Adverse Events related to the Suture-Tight Suture Delivery System | 30-days
  Recording of all Serious Adverse Event (SAE) related to the Suture-Tight™ Suture Delivery System procedure or device
Analysis of the Suture-Tight endoanchor effectiveness | 30-days
  1. Documentation of Procedural success defined as:
     * Successful delivery of the Suture-Tight™ Delivery Catheter to the site of intended treatment
     * Successful removal of Suture-Tight™ Delivery Catheter
     * Absence of evidence of acute endograft migration or dysfunction at the conclusion of the procedure
  2. Absence of a Type 1a Endo Leak
  3. Absence of a stent graft migration

SECONDARY OUTCOMES:
All cause safety events recorded during the study | 6-months
  All-cause SAEs recorded during the EVAR procedure through follow-up.
Clinical Performance of the Stent Graft following Suture-Tight implant | 6-months
  Evaluation of Changes in Stent graft patency, migration or displacement in follow-up as measured by an abdominal CT scan
Clinical Performance of the Suture-Tight following implant | 6-months
  Evaluation of the Suture-Tight™ Suture migration, displacement, or fracture as measured by an abdominal CT scan and KUB x-rays.

CONTACTS AND LOCATIONS:
Overall Officials: Ramon Varcoe, MD, Principal Investigator — Prince of Wales Private Hospital
Locations (1):
- Prince of Wales Private Hospital, Randwick, New South Wales, Australia

IPD SHARING:
Plan to Share IPD: No